CLINICAL TRIAL: NCT05111704
Title: Short-term Effects of Postural Taping on Pain and Neck Posture: a Randomized Controlled Trial
Brief Title: Short-term Effects of Postural Taping on Pain and Neck Posture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linnaeus University (Other)
Collaborators: Halmstad University (Other)
Responsible Party: Principal Investigator, Sofia Ryman Augustsson, Associate Professor, Linnaeus University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-02610
Record Dates: First submitted 2021-10-13; First posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Neck Pain, Posterior
Keywords: posture; Balance Body Tape
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: 26 subjects experiencing pain in neck, back or shoulders were randomized into either an intervention group (n=12) or control group (n=14).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balance Body Tape (Experimental): Three-week treatment with Balance Body Tape (BBT).
  Interventions: Other: Balance Body Tape
- Control group (No Intervention): Control group receiving no intervention.

INTERVENTIONS:
Other: Balance Body Tape — The intervention group received a three-week treatment with Balance Body Tape (BBT) (product by Babota AB), the control group received no treatment. A questionnaire regarding pain, including a Numeric Rating Scale (NRS) measuring pain intensity, and a Photographic posture analysis measurement (PPAM) of habitual sitting posture were accomplished before and after the intervention for both groups.
  Arms: Balance Body Tape

SUMMARY:
The aim of this study was to investigate the effects of a short treatment period with Balance Body Tape on the intensity of perceived neck, shoulder and back pain and neck posture.

DETAILED DESCRIPTION:
The aim of this study was to investigate the effects of a short treatment period with Balance Body Tape on the intensity of perceived neck, shoulder and back pain and neck posture.

Method 26 subjects who reported being university students or having a sedentary work and experiencing pain in neck, back or shoulders were randomized into intervention- (n=12) and control group (n=14).

The intervention group received a three-week treatment with BBT, the control group received no treatment. A questionnaire regarding pain, including a Numeric Rating Scale (NRS) measuring pain intensity, and a Photographic posture analysis measurement (PPAM) of habitual sitting posture were accomplished before and after the intervention for both groups. Wilcoxon´s signed rank test and Mann-Whitney U test was used to assess intra- and between group differences respectively. The relationship between pain intensity and CV-angle was assessed using Spearman's rank-order correlation.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-39
* University student or having a sedentary work
* Experienced of neck, shoulder and/or back pain, during prolonged sitting
* Minimum of 2-point score at the Numeric Rating Scale.

Exclusion Criteria:

* Severe back or neck injuries within the last 3 months
* Ongoing treatment plan for any back or neck problems
* Severe contact allergy or eczema
* Previously tried Body Balance Tape.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Three week
  Pain intensity measured by numeric rating scale (NRS) rating from 0-10, where 0=no pain and 10= worst pain
Craniovertebral angle | 6 minutes
  Neck posture measured by the craniovertebral (CV) angle in sagittal plane.

CONTACTS AND LOCATIONS:
Locations (1):
- Sofia Ryman Augustsson, Kalmar, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Augustsson SR, Reinodt S, Sunesson E, Haglund E. Short-term effects of postural taping on pain and forward head posture: a randomized controlled trial. BMC Musculoskelet Disord. 2022 Feb 19;23(1):162. doi: 10.1186/s12891-022-05083-5. PMID 35183157